CLINICAL TRIAL: NCT02128737
Title: Neurobehavioral Effects of Partial Sleep Deprivation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 810896
Record Dates: First submitted 2014-04-10; First posted 2014-05-01 (Estimated); Last update posted 2015-06-11 (Estimated); Status verified 2014-04

CONDITIONS: Control; 1 Night Recovery Sleep; 3 Nights Recovery Sleep; 5 Nights Recovery Sleep
MeSH Terms: interventions — Sleep

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control (No Intervention): 10 hours time-in-bed all nights of study
- 1 Recovery Night (Experimental): 2 baseline nights, five nights sleep restriction, 1 recovery night, five nights sleep restriction, 4 recovery nights
  Interventions: Behavioral: Sleep
- 3 Recovery Nights (Experimental): 2 baseline nights, five nights sleep restriction, 3 recovery nights, five nights sleep restriction, 2 recovery nights
  Interventions: Behavioral: Sleep
- 5 Recovery Nights (Experimental): 2 baseline nights, five nights sleep restriction, 5 recovery nights, five nights sleep restriction, 1 recovery nights
  Interventions: Behavioral: Sleep

INTERVENTIONS:
Behavioral: Sleep
  Arms: 1 Recovery Night; 3 Recovery Nights; 5 Recovery Nights

SUMMARY:
This project continues an innovative line of research on how to optimally use sleep as an intervention to promote cognitive recovery from, and resistance to, the neurobehavioral risks posed by chronic partial sleep deprivation. Chronic insufficient sleep is estimated to affect at least 20% of adults. It can result from medical conditions and sleep disorders, as well as work demands, and social or domestic responsibilities. It is associated with significant clinical morbidity, and directly causes errors and accidents that are due to its adverse neurobehavioral effects on alertness, mood, and cognitive functions. In seminal experiments conducted under this grant, we showed that the neurobehavioral effects of chronic sleep restriction accumulate to severe levels in a few days, without the full awareness of the affected individuals, and that recovery from chronic sleep restriction requires more sleep than previously assumed. We also discovered that recovery from chronic sleep was illusory, because it masked a heightened neurobehavioral vulnerability to even a single post-recovery night of sleep restriction. The implications of these findings are that apparent recovery from chronic sleep restriction masks a more severe cognitive response to subsequent sleep restriction suggesting that there are longer time constants in the brain for neurobehavioral recovery from chronic sleep restriction. In light of this finding, we now seek to determine whether additional nights of extended recovery sleep will reduce the heightened vulnerability induced by prior exposure to sleep restriction. A total of 87 healthy adults (ages 21-50) will be studied in the laboratory during a 17-night (N=63) and a 19-night (N=24) protocol evaluating cognitive, psychological and physiological responses to varying recovery days between two sleep-restriction periods. The results will establish the number of nights of recovery sleep needed to prevent accelerated deterioration during a subsequent period of sleep restriction. The findings will advance theoretical understanding of sleep homeostasis and its relationship to cognitive functions, as well as inform theories of sleep need, and have substantial implications for sleep biology, for the treatment of clinical disorders that regularly disrupt sleep, and for managing lifestyle factors that frequently restrict sleep.

ELIGIBILITY:
Inclusion Criteria:

A total of N=87 adult subjects (aged 21-50 yr), N=43 females and N=44 males of all ethnicities, will be randomized to the 3 different conditions (n=26 for each of 2 experimental conditions; n=11 for the control condition) for the 17-night protocol or assigned to the 5-night experimental recovery condition (n=24) for the 19-night protocol. Subjects must also be comparable in terms of their homeostatic and circadian sleep-wake regulation parameters. In order to be eligible to participate, subjects must meet the following inclusion criteria:

1. Age between 21 and 50 years (average age of our current protocols is 31 years)
2. Body mass index (BMI) within 20.5% of normal
3. Stable, normally-timed sleep-wake cycle as determined by interview, 2-week daily sleep log, and 2-week wrist actigraphic evidence, and defined by:
4. Habitual nocturnal sleep duration between 6.5h and 8.5h
5. Habitual morning awakening between 0600h and 0930h

Exclusion Criteria:

1. No evidence of habitual napping
2. No shift work, transmeridian travel or irregular sleep/wake routine in the past 60 days
3. No sleep disorder, determined by history, actigraph, pulse oximetry and PSG
4. No history of mania or psychosis
5. No current depression as determined by the Beck Depression Inventory
6. No alcohol or drug abuse in the past year based upon history and urine toxicology screen
7. Not a current smoker
8. No acute, chronic, or debilitating medical conditions, major Axis I psychiatric illness, epilepsy, or thyroid disease, based on history, physical exam, blood and urine chemistries, and CBC

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2009-12; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Psychomotor Vigilance Test | Assessed everyday of the in-laboratory study (17 days) and is completed every 2 hours
  3, 10 or 20 minute simple, high-signal-load reaction time (RT)-based test invented by our group and designed to evaluate the ability to sustain attention and respond in a timely manner to salient signals.

CONTACTS AND LOCATIONS:
Overall Officials: David F Dinges, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- Unit for Experimental Psychiatry, Sleep and Chronobiology Laboratory, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Spaeth AM, Dinges DF, Goel N. Objective Measurements of Energy Balance Are Associated With Sleep Architecture in Healthy Adults. Sleep. 2017 Jan 1;40(1):zsw018. doi: 10.1093/sleep/zsw018. PMID 28364451
- [Derived] Spaeth AM, Dinges DF, Goel N. Sex and race differences in caloric intake during sleep restriction in healthy adults. Am J Clin Nutr. 2014 Aug;100(2):559-66. doi: 10.3945/ajcn.114.086579. Epub 2014 Jun 25. PMID 24965304